CLINICAL TRIAL: NCT06546696
Title: The ADAPT Trial: Adapting Evidence-Based Obesity Interventions in Community Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Bill Heerman, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 241092
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This is cluster-randomized trial, where we anticipate randomizing 50 community centers and enrolling 750 children (15/center).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COACH Intervention (Experimental): COACH intervenes at 3 levels: the individual child, the family, and the community.
  Child-Level Intervention Content: We will direct skill-building lessons toward the child at developmentally appropriate levels.
  Family-Level Intervention Content: Curricular components for parents are designed to leverage parents as agents of change for their children. As such, the group-based sessions includes realistic goal setting (SMART goals), strategies to navigate barriers, training in physical activity, and group-based accountability. During the session, parents and children will participate in a low to moderate physical activity.
  Community-Level Content: The intervention is delivered in the context of a widely available community resource, local community centers across Middle Tennessee.
  Online Platform: All participants will have access to an online on-demand health behavior change curriculum. Modules are self-paced and will take approximately 7 hours.
  Interventions: Behavioral: Competency Based Approaches to Community Health (COACH)
- Adaptation Arm (Active Comparator): The core components of the adaptation arm will mirror the COACH intervention arm. Each community center will be guided through a process of adapting the specific intervention content, and as such, will be unique to each of the 25 community centers randomized to this arm. In this way, the study tests the process of adapting the intervention, instead of a specific portfolio of adaptations.
  Interventions: Behavioral: Competency Based Approaches to Community Health (COACH)

INTERVENTIONS:
Behavioral: Competency Based Approaches to Community Health (COACH) — COACH is a multi-level intervention, consisting of 1) developmentally appropriate health curriculum for children; 2) family-based content that both targets parent weight loss and leverages a shared parent-child experience to improve family health behaviors; 3) community-level intervention to improve access and quality of family-based programming at local Parks and Rec centers.
  Other Names: COACH

SUMMARY:
Evidence-based obesity treatment is inaccessible to most children in the United States. This lack of access is a source of health inequity, whereby children from rural and minority communities, who have the highest rates of childhood obesity, are also the least likely to receive an evidence-based intervention. Developing strategies to improve access to evidence-based obesity interventions could reduce health disparities by improving reach to these underserved communities. The premise of this study is that using a systematic framework to adapt a community-based behavioral intervention for childhood obesity that accounts for individual, family, and community factors will increase reach and effectiveness among low-income, minority, and rural populations. COACH is a multi-level obesity intervention that supports 1) the individual child through developmentally appropriate health behavior curriculum, 2) the family by directly addressing parent weight loss and engaging parents as agents of change for their children, and 3) the community by building the capacity of local community centers to offer parent-child programming. The investigators propose testing the process of adapting COACH in a cluster-randomized trial.

DETAILED DESCRIPTION:
In Aim 1, the investigators will conduct a community readiness assessment for COACH in 50 community centers serving rural, minority, and low-income families in middle TN. In 25 randomly selected community centers, the investigators will use a systematic process to adapt the intervention protocol based on the assessment results, while maintaining fidelity to COACH's core components. In Aim 2, in a cluster-randomized trial, the investigators will test the comparative effectiveness of each implementation strategy (adaptation vs. original program) on the implementation outcomes of reach, adoption, implementation, and maintenance. In Aim 3, the investigators will test the comparative effectiveness of the adapted and original intervention.

This research is innovative because it uses adaptation science as a potential solution to reduce health disparities in childhood obesity. By testing this intervention in a community resource available to 230 million Americans (community centers), the investigators aim to create a scalable obesity intervention that could be implemented in traditionally underserved populations across the country. This study will also develop and test a theory-based process for adapting behavioral interventions for both obesity and other health outcomes among diverse rural and urban communities.

ELIGIBILITY:
Inclusion Criteria:

* Child with an age ≥ 6 years and < 12 years
* Child body mass index ≥95th percentile for age and sex on standardized CDC growth curves
* Index parent/legal guardian with an age ≥18 years
* Parent and child speak English or Spanish
* Family resides within or frequently visit selected zip codes within Middle TN surrounding the partnering community centers;
* Have parental commitment to participate in a 6-month study;
* Have the ability to view online trainings
* Complete baseline data collection, including parent and child height and weight and at least 90% of baseline survey items.

Exclusion Criteria:

* Participant child has been diagnosed with Down Syndrome, Autism, or any other developmental disorders that impact metabolism or behaviors that would preclude participation in group physical activity settings;
* Either the participant caregiver or child is unable to participate in light to moderate physical activity;
* Participant caregiver has a serious mental or neurologic illness that impairs ability to consent/participate.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Child Percent of the 95th Body Mass Index Percentile | 6 months post randomization
  Calculated from CDC growth curves

SECONDARY OUTCOMES:
Child Percent of the 95th Body Mass Index Percentile | 6 weeks post randomization
  Calculated from CDC growth curves

OTHER OUTCOMES:
Child Diet | 6 months post randomization
  Child Nutrition and Physical Activity Behavior Scale. Possible range of 0-9 with higher scores indicating healthier diet and physical activity practices.
Child Physical Activity | 6 months post randomization
  Child Nutrition and Physical Activity Behavior Scale. Possible range of 0-9 with higher scores indicating healthier diet and physical activity practices.
Child Media Use | 6 months post randomization
  Child Media Use Index
Child Sleep | 6 months post randomization
  Children's Sleep Habits Questionnaire
Parent Body Mass Index | 6 weeks post randomization
  Measured by study staff
Parent Body Mass Index | 6 months post randomization
  Measured by study staff

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Following the study's conclusion, aggregate data may be made available based on reasonable request.
  We will plan to upload a de-identified dataset to the NHLBI BioLINCC database (this upload also includes study protocols).